CLINICAL TRIAL: NCT06297135
Title: Loving Habits: A Feasibility Study of a Support Program for Building New Parent-child Behavioral Habits
Brief Title: A Feasibility Study of a Support Program for Building New Parent-child Behavioral Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okinawa Institute of Science and Technology Graduate University (Other)
Collaborators: Miyazaki International College (Other); Japan society for the promotion of science (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR-2023-020
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral intervention group (Experimental): Parents who enroll in the program will receive a series of 6 videos (~7 minutes each), 1 video at a time, generally every 3 days. Parents will also receive daily written texts, which include implementation tips and an assessment of a target (transition) behavior.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Teaches parents antecedent- and reinforcement-based behavior management techniques and provide support to manage their stress

SUMMARY:
This study evaluates the feasibility and preliminary impacts of a new parent support program consisting of a series of educational videos, delivered via a popular texting platform. For this pilot project, the program content is focused on teaching parents strategies to better manage one of the commonly reported challenges children face, a transition to a non-preferred activity. Parents with children demonstrating inattentive, hyperactive and impulsive behavior and experiencing difficulties with daily transition routines are invited to participate in the study.

DETAILED DESCRIPTION:
This pilot study employs a pre-post, open trial design with the primary aim to investigate the feasibility of delivering parenting educational materials in an accessible format, i.e., a widely used testing platform. The training videos demonstrate the applications of antecedent- and reinforcement-based behavior management techniques in a specific situation and encourage parents to build positive parenting habits. The program usability and satisfaction will be assessed through participant ratings. The study targets parents of children demonstrating inattention, hyperactive, and impulsive behavior. These families frequently experience difficulties managing everyday routines at home, yet the access to psychosocial treatment is limited. The investigators expect parents to engage well in the program delivered via digital media. Based on the existing literature on the effectiveness of behavior parent training delivered in traditional in-person format, a moderate effect size is expected in the pre-post measures of parenting practices and the child target behavior for this study.

ELIGIBILITY:
Inclusion Criteria:

Parents with children aged 4-10, who experience difficulties with transitions. The program will be advertised that it was developed targeting children demonstrating behaviors consistent with ADHD, and the ADHD symptoms will be measured pre-post. However, children are not required to have a diagnosis of ADHD or show elevated levels of ADHD symptoms for the parents to sign up.

Exclusion Criteria:

Parents who do not understand Japanese (the language the program is offered in).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number of videos viewed | 1 month
  The number of videos viewed (minimum 0, maximum 6) to evaluate participant engagement.
Percentage of completed daily ratings | 1 month
  The percentage of completed daily ratings (minimum 0, maximum 100). Parents are asked to provide daily ratings on the degree of success in implementing parenting strategies taught.
Participant satisfaction | 1 month
  The parent-rated satisfaction regarding information presented in the videos. A rating completed after each video viewing using a 4-point scale. Averaged across the ratings completed for the videos viewed. (Minimum 0, maximum 4). Higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Parent-rated child's difficulties with daily transitions | 1 month
  The parent-rated child's difficulties with 9 common daily transitions. Ratings completed before and after the intervention using a 3-point scale. Averaged across the ratings completed for the 9 transitions. Higher scores indicate greater difficulties.
Parent-rated child's impairment related to transition difficulties | 1 month
  The parent-rated level of impairment caused by transition difficulties (1 item). Ratings completed before and after the intervention using a 7 point scale. Higher scores indicate greater impairment.
Positive parenting | 1 month
  Positive and Negative Parenting Scale (PNPS) Positive Parenting sub-scale. Parent ratings completed before and after the intervention using a 4-point scale. Average across 8 items. Higher scores indicate more frequent use of positive parenting strategies.
Negative parenting | 1 month
  Positive and Negative Parenting Scale (PNPS) Negative Parenting sub-scale. Parent ratings completed before and after the intervention using a 4-point scale. Average across 8 items. Higher scores indicate more frequent use of negative parenting strategies.
Parenting stress | 1 month
  Parent Stress Scale total score. Parent ratings completed before and after the intervention using a 5-point scale. Average across 18 items. Higher scores indicate higher levels of parent stress.

OTHER OUTCOMES:
ADHD symptoms | 1 month
  SNAP-IV inattention and hyperactivity/impulsivity symptoms total. Parent ratings completed before and after the intervention using a 4-point scale. Averaged across 18 items. Higher scores indicate ADHD symptoms more frequently observed.
ODD symptoms | 1 month
  SNAP-IV oppositional/defiant symptoms total. Parent ratings completed before and after the intervention using a 4-point scale. Averaged across 8 items. Higher scores indicate ADHD symptoms more frequently observed.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Miyazaki International College, Miyazaki, Miyazaki
  - Okinawa Institute of Science and Technology Graduate University, Onna, Okinawa

IPD SHARING:
Plan to Share IPD: No